CLINICAL TRIAL: NCT01305681
Title: Bacterial Properties With LoFric® Catheters During Clean Intermittent Catheterization
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: It appears Dr. Vanderbrink left Nationwide Children's Hospital in 2011 and efforts to reach Dr. Vanderbrink have been unsuccessful.
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB10-00458
Record Dates: First submitted 2011-02-28; First posted 2011-03-01 (Estimated); Last update posted 2019-08-07 (Actual); Status verified 2011-11

CONDITIONS: Neurogenic Bladder; Urinary Retention
MeSH Terms: conditions — Urinary Bladder, Neurogenic; Urinary Retention

STUDY DESIGN:
Intervention Model Description: It appears Dr. Vanderbrink left Nationwide Children's Hospital in 2011 and efforts to reach Dr. Vanderbrink have been unsuccessful. The study expired with the NCH IRB before it was ever approved for a 2nd year.
Masking Description: Please close this study at ct.gov as we have not further data at NCH as Dr. Vanderbrink left NCH in 2011.

ARMS (1):
- LoFric® catheters (Active Comparator): LoFric® catheters during clean intermittent catheterization will be compared to non-LoFric® catheters during clean intermittent catheterization
  Interventions: Device: LoFric® catheters during clean intermittent catheterization

INTERVENTIONS:
Device: LoFric® catheters during clean intermittent catheterization — LoFric® catheters during clean intermittent catheterization

SUMMARY:
The primary objective of our study is to examine characteristics of bacteria that are discovered in urine from pediatric patients that utilize either LoFric® or non-LoFric® catheters for self intermittent catheterization. The investigators hypothesize that the hydrophilic nature of the LoFric® catheter will alter the microbial environment and reduce clinically significant urinary tract infections in patients with neurogenic bladder compared to a similar population using standard catheters.

Secondary outcomes will be comparing the incidence of clinical urinary tract infections between patients that use standard catheters and those that use LoFric catheters.

Lastly, patient satisfaction using LoFric catheters compared to standard catheters will be assessed.

DETAILED DESCRIPTION:
The investigators will randomize patients with neurogenic bladder into 2 groups after the have been matched for age, gender and mobility.

The first group will continue with their current intermittent catheterization system (a non-LoFric® catheter) while the second group will receive sufficient LoFric® catheters to complete the study. The investigators will collect the urine at the start of the study, and then at 3, 6, 12, and 18 months and sent for culture. If a child develops a urinary tract infection, the investigators will have the patient collect the urine and the urine will be cultured and the organism will be identified.

Using an existing bladder cell line, the investigators will inoculate the bladder cells with any bacteria that grows from any sample and then determine the interleukin-6 response of the bladder cell line following inoculation with the bacteria. This will determine if the initiate a high or low cytokine response which the investigators have correlated to clinical risk of symptomatic urinary tract infection

The investigators will provide a patient satisfaction survey at the start of the study, prior to randomization and at the completion of the study to determine satisfaction with LoFric® catheters.

ELIGIBILITY:
Inclusion Criteria:

* Patients who perform clean intermittent catheterization on a regular basis

Exclusion Criteria:

* Patients on daily continuous antibiotic therapy

Max Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2011-05-06 (Actual); Primary Completion 2012-02-21 (Actual); Study Completion 2012-02-21 (Actual)

PRIMARY OUTCOMES:
Characteristics of bacteria discovered in urine of pediatric patients using LoFric® catheters during clean intermittent catheterization | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States